CLINICAL TRIAL: NCT04827082
Title: Effects of Diacutaneous Fibrolysis on Flexibility and Active Neuromuscular Response on Posterior Muscular Chain of Lower Limb in Athletes
Brief Title: Effects of Diacutaneous Fibrolysis on Flexibility and Active Neuromuscular Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Aida Cadellans Arróniz, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIS202004
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Hamstring Contractures
Keywords: Diacutaneous fibrolysis; Physiotherapy; Neuromuscular response

STUDY DESIGN:
Intervention Model Description: A randomized control trial
Who Masked: Outcomes Assessor
Masking Description: The assessor will not know if patient have received the treatment or not
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diacutaneous fibrolysis group (Experimental): Diacutaneous fibrolysis is a physiotherapeutic instrumental technique, used to treat musculoskeletal conditions causing pain and/or movement restriction. It is applied by means of metallic hooks, ending in a spatula with beveled edges. Regardless of its own dominance, diacutaneous fibrolysis will be applied to de following muscles and intermuscular septums: gluteus maximus, biceps femoris and semitendinosus to de lower experimental limb. A single session of 10 minutes will be applied.
  Interventions: Other: Diacutaneous fibrolysis
- Control group (No Intervention): Participants will be used as their own controls, with one lower extremity randomly receiving intervention. The control extremity will not receive any intervention

INTERVENTIONS:
Other: Diacutaneous fibrolysis — Diacutaneous fibrolysis is a physiotherapeutic instrumental technique, used to treat musculoskeletal conditions causing pain and/or movement restriction. It is applied by means of metallic hooks, ending in a spatula with beveled edges. Regardless of its own dominance, diacutaneous fibrolysis will be applied to de following muscles and intermuscular septums: gluteus maximus, biceps femoris and semitendinosus to de lower experimental limb. A single session of 10 minutes will be applied.
  Arms: Diacutaneous fibrolysis group

SUMMARY:
Diacutaneous fibrolysis is a physiotherapeutic instrumental technique, used to treat musculoskeletal conditions causing pain and/or movement restriction. It is applied by means of metallic hooks, ending in a spatula with beveled edges, that seems to allow a better pressure distribution on the skin and a deeper and more precise application, compared to the manual approach. Recent studies indicate positive responses regrading pain intensity decrease in sports people suffering anterior knee pain, improving range of motion in subacromial impingement syndrome, improving sensory conductivity in symptomatic patients with carpal tunnel syndrome, decreased pain in patients with chronic epicondialgia or improveing function athletes with anterior knee pain. However, the specific action mechanism, have not been investigated in depth yet. There are no studies evaluating its effects on posterior muscular chain of lower extremity in athletes, where FD effects on neuromuscular response could be more evident due to the overload involved on this area. The aim of this study is to evaluate the immediate, and after 30 minutes, effects of a single diacutaneous fibrolysis session on flexibility, strength and neuromuscular activity on hamstring in athletes. A randomized controlled trial with blind evaluator. Randomization will be done between lower extremities of each subject (Random.org). Regardless of its own dominance, diacutaneous fibrolysis will be applied to de following muscles and intermuscular septums: gluteus maixmus, biceps femoris and semitendinosus to de lower experimental limb. The other extremity will not be treat (control limb).

Sample recruitment. Athletes from UIC university community, who compete officially or institutionally, whether they are federated or recorded in a sport official register where the predominant activity focuses on the lower train (athletics, cycling, football, rugby...). Procedure. The anthropometric data will be collected at the beginning of the study. Each outcome assessment will be performed by a blinded evaluator at the baseline, immediately after the technique application and 30 minutes after.

ELIGIBILITY:
Inclusion Criteria:

* Athletes
* <160º in the Passive Knee Extension test
* Participants must sign and have informed consent.

Exclusion Criteria:

* Poor skin
* Trophic condition
* Taking anticoagulants
* Inflammatory process
* Recent musculoskeletal lower limb injury (< 6 month)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Hamstring neuromuscular activity | Change between baseline (immediately before intervention) and post intervention (immediately after intervention); Change between baseline (immediately before intervention) and 30 minutes after intervention]
  Hamstring neuromuscular activity (% of muscular fiber recruitment) will be assessed by surface electromyogram (mDurance). The electrodes will be placed on hamstring muscle while performing a functional movement.
Gluteus maximus neuromuscular activity | Change between baseline (immediately before intervention) and post intervention (immediately after intervention); Change between baseline (immediately before intervention) and 30 minutes after intervention]
  Gluteus maximus neuromuscular activity (% of muscular fiber recruitment) will be assessed by surface electromyogram (mDurance). The electrodes will be placed on gluteus maximus muscle while performing a functional movement.
Hamstring isometric strength | Change between baseline (immediately before intervention) and post intervention (immediately after intervention); Change between baseline (immediately before intervention) and 30 minutes after intervention]
  Isometric muscle strength (Kg) will be evaluated by means of a digital dynamometer (Microfeet 2). This measures will be taken across a knee flexion.
Guteus maximus isometric strength | Change between baseline (immediately before intervention) and post intervention (immediately after intervention); Change between baseline (immediately before intervention) and 30 minutes after intervention]
  Isometric muscle strength (Kg) will be evaluated by means of a digital dynamometer (Microfeet 2). This measures will be measured by means of hip extension.
Height on counter movement jump | Change between baseline (immediately before intervention) and post intervention (immediately after intervention); Change between baseline (immediately before intervention) and 30 minutes after intervention]
  Height (centimeters) on counter movement jump will be assessed using a mobile application called "My jump". Its data has been used as an indirect indicator of explosive muscular strength of lower limb
Time flight on counter movement jump | Change between baseline (immediately before intervention) and post intervention (immediately after intervention); Change between baseline (immediately before intervention) and 30 minutes after intervention]
  Time flight (milliseconds) on counter movement jump will be assessed using a mobile application called "My jump".
Force on counter movement jump | Change between baseline (immediately before intervention) and post intervention (immediately after intervention); Change between baseline (immediately before intervention) and 30 minutes after intervention]
  Force (newtons) on counter movement jump will be assessed using a mobile application called "My jump".
Back chain flexibility Changes | Change between baseline (immediately before intervention) and post intervention (immediately after intervention); Change between baseline (immediately before intervention) and 30 minutes after intervention]
  Back chain flexibility is going to be assessed by means of modified Back Saver Sit and reach test (centimeters).
Hamstring flexibility changes | Change between baseline (immediately before intervention) and post intervention (immediately after intervention); Change between baseline (immediately before intervention) and 30 minutes after intervention]
  Hamstring muscles flexibility will be assessed using the passive knee extension test (degrees) by means of goniometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided